CLINICAL TRIAL: NCT07392567
Title: A Multicenter, Prospective, Observational Study for the Validation of a Multimodal Deep Learning Model to Predict Metachronous Liver Metastasis in Patients With Colorectal Cancer After Curative Resection
Brief Title: Prospective Validation of an AI Model for Predicting Liver Metastasis in Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Prof., Tongji Hospital
Other Study IDs: TJ-IRB202601017
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Liver Metastasis
Keywords: colorectal cancer liver metastasis; deep learning; multimodal; predictive model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Validation Cohort: This single cohort consists of patients with stage I-III colorectal cancer who are prospectively enrolled after undergoing curative resection. No interventions are administered as part of this study. The cohort is used for the external validation of the pre-defined multimodal deep learning model's performance in predicting the risk of metachronous liver metastasis. All patients receive standard of care treatment and follow-up according to clinical guidelines.
  Interventions: Diagnostic Test: Multimodal Deep Learning Prediction Model

INTERVENTIONS:
Diagnostic Test: Multimodal Deep Learning Prediction Model — This is a non-therapeutic, prognostic study. The intervention under investigation is the application of a pre-specified multimodal deep learning model that integrates preoperative CT imaging, digital pathology, and clinical data to stratify patients' risk of developing metachronous liver metastasis. This model functions as a prognostic tool and is not used to guide patient management in this study. Its performance is being evaluated prospectively against the actual clinical outcomes.

SUMMARY:
This is a prospective, multicenter, observational study designed to validate the predictive accuracy of a pre-developed multimodal deep learning model. The model integrates preoperative contrast-enhanced CT scans, digitized postoperative pathology images, and standard clinical data to estimate the risk of liver metastasis within two years after curative surgery in patients with stage I-III colorectal cancer.

The primary objective is to evaluate the model's performance in an independent, prospectively enrolled patient cohort. Participants will receive standard-of-care treatment according to clinical guidelines. The study involves no experimental interventions; it solely involves the collection and analysis of routinely generated clinical data. The goal is to assess the model's potential for clinical translation by providing a reliable tool for stratifying patients' risk of liver metastasis, which could inform personalized surveillance strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, any gender.
* Clinical diagnosis of primary colon or rectal adenocarcinoma (Stage I-III). Scheduled to undergo curative radical resection for colorectal cancer.
* Preoperative contrast-enhanced abdominal/pelvic CT scan performed within 1 month before surgery, with acceptable image quality.
* No evidence of distant metastasis (including synchronous liver metastasis) on preoperative examination.
* ECOG Performance Status of 0 or 1.
* Patient or their legal representative voluntarily participates and provides written informed consent.

Exclusion Criteria:

* Postoperative pathological confirmation of non-primary colorectal adenocarcinoma or presence of distant metastasis.
* Intraoperative determination of non-R0 resection, or performance of palliative surgery/ostomy only.
* History of other malignant tumors.
* Previous history of liver surgery or liver transplantation.
* Death within the perioperative period (within 30 days after surgery).
* Refusal to participate in follow-up, withdrawal of informed consent, or loss to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population consists of adult patients (aged 18-75) with newly diagnosed, stage I-III primary colorectal cancer who are scheduled to undergo curative resection at one of the participating clinical centers. This prospective cohort will be used for the independent validation of a pre-developed multimodal deep learning model designed to predict the risk of metachronous liver metastasis. All participants will provide informed consent prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) | 2 years after surgery
  The discriminatory performance of the pre-specified multimodal deep learning model for predicting the occurrence of metachronous liver metastasis within 2 years after curative resection. The model integrates preoperative contrast-enhanced CT, digital pathology, and clinical data. Performance is evaluated on the entire prospectively enrolled validation cohort.

SECONDARY OUTCOMES:
Liver Metastasis-Free Survival (LMFS) by Risk Group | From the date of surgery until the date of first documented liver metastasis or last follow-up, assessed up to 3 years.
  The difference in liver metastasis-free survival between the high-risk and low-risk groups, as stratified by the model. LMFS is defined as the time from surgery to the first radiological diagnosis of liver metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No